CLINICAL TRIAL: NCT03946215
Title: Comparison of Cardiorespiratory Responses to Treadmill Running at Different Slopes in Well-trained Athletes
Brief Title: Cardiorespiratory Responses to Treadmill Running at Different Slopes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 7038
Record Dates: First submitted 2018-08-31; First posted 2019-05-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cardiorespiratory Responses; Well-trained Athletes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- well-trained athletes (Experimental): A cardiorespiratory stress test
  Interventions: Other: Each participant will perform:

INTERVENTIONS:
Other: Each participant will perform: — Part 1: Maximal incremental tests will require running at fixed slopes (+15%, 0% -15%) for stages (2min duration) of increasing velocities (0.5, 1 and 1.5 km/h) Part two: submaximal running tests will require running at constant velocity (80% VO2max uphill; 80%VO2max downhill and downhill at similar velocity as uphill)

SUMMARY:
The purpose of this study is: i) to determine if maximal oxygen uptake in downhill running is significantly different versus flat or uphill running, and ii) to compare cardiorespiratory and muscle fatigue responses to uphill vs flat and downhill running at similar running velocity and similar metabolic power. The investigators hypothesized that maximal oxygen uptake will be lower in downhill running. The investigators also anticipate attenuated cardiorespiratory and muscle fatigue responses to downhill running when compared to flat or uphill running performed at similar velocity but not when the comparison is done at similar metabolic power.

ELIGIBILITY:
Inclusion Criteria:

* to be a well-trained runner with a VO2max > à 55 ml/kg/min
* nonsmoker or stopped smoking for 5 years
* BMI < 25
* affiliation to the social health insurance scheme
* signing an informed consent form.

Exclusion criteria:

* impossibility to give the subject enlightened information (subject in emergency situation, difficulties in understanding the study, ...);
* subject under the protection of justice
* subject under guardianship or curatorship
* contraindication to the practice of physical and sport activities
* lower limbs musculotendinous or articular problems
* respiratory, cardiovascular or metabolic pathology
* drug treatment in progress and impossibility to stop it within 7 days before the beginning of the study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Peak oxygen | 15 minutes
  The peak oxygen uptake will be collected during downhill, flat and uphill running

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lemire M, Hureau TJ, Remetter R, Geny B, Kouassi BYL, Lonsdorfer E, Isner-Horobeti ME, Favret F, Dufour SP. Trail Runners Cannot Reach V O2max during a Maximal Incremental Downhill Test. Med Sci Sports Exerc. 2020 May;52(5):1135-1143. doi: 10.1249/MSS.0000000000002240. PMID 31815832